CLINICAL TRIAL: NCT06790862
Title: A Multicenter, Randomized, Double-blind, Parallel, Excipient-controlled Phase II Clinical Study Evaluating the Efficacy and Safety of SHR0302Base in Subjects With Nonsegmental Vitiligo
Brief Title: A Trial of SHR0302Base in Patients With Vitiligo
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR0302Base-201
Record Dates: First submitted 2025-01-20; First posted 2025-01-24 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Intervention Model Description: SHR0302Base compared with placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Treatment group 1 (Experimental)
  Interventions: Drug: SHR0302Base gel
- Treatment group 2 (Experimental)
  Interventions: Drug: SHR0302Base gel
- Treatment group 3 (Experimental)
  Interventions: Drug: SHR0302Base gel
- Treatment group 4 (Placebo Comparator)
  Interventions: Drug: SHR0302Base gel placebo

INTERVENTIONS:
Drug: SHR0302Base gel — SHR0302Base gel.
  Arms: Treatment group 1; Treatment group 2; Treatment group 3
Drug: SHR0302Base gel placebo — SHR0302Base gel placebo.
  Arms: Treatment group 4

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of SHR0302Base in participants with nonsegmental vitiligo.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically diagnosis of non-segmental vitiligo.
2. The disease has been stable for more than 3 months (90 days) (stable disease is defined as no expansion of the original lesion and no new lesions).
3. Subjects and their partners do not plan to have children, do not donate sperm/eggs, and voluntarily use highly effective contraception during the study period until 6 months (female subjects) or 3 months (male subjects) after dosing. Female subjects must have a negative serum pregnancy test and be non-lactating.

Exclusion Criteria:

1. Subjects diagnosed with segmental, mixed or undifferentiated vitiligo; Or previously diagnosed with other skin pigmentation disorders (except nevus halos).
2. Conditions at baseline that would interfere with evaluation of vitiligo.
3. Participants who have used skin bleaching treatments for past treatment of vitiligo or other pigmented areas.
4. Use of protocol-defined treatments within the indicated washout period before baseline.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2025-02-13 (Actual); Primary Completion 2026-03-03 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects who achieved at least a 50% improvement from baseline in the facial-neck vitiligo area score (F-VASI 50 response). | At week 24.

SECONDARY OUTCOMES:
The proportion of subjects who achieved at least a 75% improvement from baseline in the facial-neck vitiligo area score (F-VASI 75 response). | At week 24.
The proportion of subjects who achieved at least a 90% improvement from baseline in the facial-neck vitiligo area score (F-VASI 90 response). | At week 24.
The proportion of subjects who achieved at least a 50% improvement from baseline in the overall vitiligo area score index from baseline (T-VASI 50 response). | At week 24.
The proportion of subjects who achieved at least a 75% improvement from baseline in the overall vitiligo area score index from baseline (T-VASI 75 response). | At week 24.
The proportion of subjects who achieved at least a 90% improvement from baseline in the overall vitiligo area score index from baseline (T-VASI 90 response). | At week 24.

CONTACTS AND LOCATIONS:
Locations (1):
- Dermatology Hospital affiliated to Shandong First Medical University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided